CLINICAL TRIAL: NCT04181320
Title: Multicentre, Prospective, Randomized, Open-label, Assessor Blinded Study to Evaluate Granulox® Used as Adjunct Therapy to Defined Standard of Care vs. Defined Standard of Care for the Treatment of Predominantly Chronic Venous Leg Ulcers (VLUs)
Brief Title: A Multicentre European Study to Evaluate Granulox® Used in the Treatment Pathway of Predominantly Chronic Venous Leg Ulcers (VLUs).
Acronym: Granulox01
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results of interim analysis
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Granulox01 (PD-568268)
Record Dates: First submitted 2019-11-22; First posted 2019-11-29 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-08

CONDITIONS: Venous Leg Ulcer
Keywords: Granulox; venous ulcers; wound healing; wound reduction
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: Multicentre, prospective, randomized, European open label, assessor blinded, 2-arm parallel group study.
Who Masked: Outcomes Assessor
Masking Description: Wound closure (CCC and PCC) will be assessed through ulcer photos by 2 independent and experienced clinicians unaware of treatment allocation (blind review).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venous Leg Ulcer Standard of Care (No Intervention): Subjects will recieve standard of care treatment.
- Venous Leg Ulcer Standard of Care with Granulox (Experimental): Subjects will recieve standard of care treatment with Granulox added as an adjunct therapy.
  Interventions: Device: Venous Leg Ulcer Standard of Care with Granulox

INTERVENTIONS:
Device: Venous Leg Ulcer Standard of Care with Granulox — Granulox will be added as an adjunct therapy to defined standard of care in subjects with predominantly venous leg ulcers.
  Other Names: Granulox
  Arms: Venous Leg Ulcer Standard of Care with Granulox

SUMMARY:
The investigation is designed as an open label, randomized, prospective, assessor blinded, multi centre investigation.

254 evaluable subjects will be randomized to either standard of care group or standard of care with Granulox added as an adjunct therapy in predominantly venous leg ulcer subjects. Standard of care wound management will be completed, including wound cleansing, debridement if necessary and application of a suitable dressing and compression system until complete wound closure.

The study will be divided into two phases. Firstly, a two week run-in period to ensure compliance to compression therapy followed by a 20 weeks treatment period starting with randomization and allocation of treatment.

DETAILED DESCRIPTION:
The current study is designed to verify previous clinical findings and to pinpoint clinically relevant efficacy, associated to intended use of Granulox® as a therapy added to a defined standard of care in the management of chronic VLUs. The most relevant outcome is considered to be an increase in healing of chronic VLUs over a period of 20 weeks.

This is a multi-centre European open label randomised 2-arm parallel group study. The study will include multiple European counties (e.g. France, Germany, UK, Poland, Croatia and Czech Republic), with approximately 2-7 clinics per country.

The study will run with a two-phase set-up, with a 14 days run-in period and a an up to 20 weeks treatment period starting with randomization and allocation of treatment. Confirmation of wound closure is further assessed after a 15 day followup period.

The primary objective of the study is to compare wound healing between management of chronic VLUs with or without added Granulox®. The main efficacy criterion is Confirmed Complete wound Closure (CCC).

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent to participate.
2. No planned hospitalization in the forthcoming 20 weeks.
3. Male or female (women of childbearing age must have an acceptable method of birth control).
4. Age >18 years.
5. Recent (less than 12 months) doppler or duplex colour ultrasonography compatible with chronic venous insufficiency.
6. ABPI (less than 3 months) ≥0.7 for both legs. If ABPI >1.4, then big toe pressure >60mmHg is required or an alternative measurement verifying normal distal arterial flow.
7. At least one or more supra- or peri-malleolar leg ulcers and no foot ulcer or another chronic wound.
8. In case of two or more ulcers, select ulcer with the highest PUSH score at randomization and treat the non-selected ulcer in the same way as ulcers in the control group (standard of care).
9. In case of two or more ulcers on the same limb, ensure that the distance between each ulcer is 3 cm as measured from the margins of each ulcer that are closest to one another.
10. Wound duration ≥ 8 weeks and ≤60 months.
11. At randomization, the ulcer area should be 3 cm2 - 70 cm² and should not have decreased by more than 30% during the 2-week run-in period.
12. Less than 50% of the wound area should be covered with fibrinous tissue at randomization and after debridement.
13. Patients considered as compliant/adherent to the compression device during the run-in period (i.e. no more than 2 days without compression over the 2-week run-in period).
14. No clinically significant comorbidities requiring the use of systemic steroids or any cytotoxic or immunosuppressive agents.

Exclusion Criteria:

1. Infected ulcer according to the judgment of the investigator defined as any wound condition requiring the prescription or continuation of systemic antibiotic therapy at randomization.
2. Circumferential wounds.
3. Wound covered fully or partially by necrotic tissue (black tissue).
4. Patients who will have problems following the protocol, especially compression therapy.
5. Patients included in another on-going clinical investigation, or patients who have participated in a clinical investigation during the past 30 days.
6. Wounds treated with dressings containing an active component (e.g. silver, nanooligosaccharide factor (NOSF), charcoal, chlorhexidine, iodine or ibuprofen) 14 days prior to study enrollment.
7. Patient with a systemic infection not controlled by suitable antibiotic treatment.
8. Current treatment with radiotherapy, chemotherapy, immunosuppressant drugs or high doses of oral corticosteroids (>10 mg Predinsolone or equivalent) if any.
9. Patient with deep vein thrombosis within 3 months prior to inclusion.
10. Known allergy/hypersensitivity to the ingredients of the dressings and/or Granulox®.
11. Malignant wounds.
12. Endovenous surgery planned or performed within the past 30 days.
13. Primary lymphoedema caused by congenital/developmental defect, i.e. Milroy's disease (congenital lymphedema), Meige's disease (lymphedema praecox), or Late-onset lymphedema (lymphedema tarda).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Dissemond, Professor Dr., Principal Investigator — University Hospital, Essen
Locations (27):
- Croatia (3):
  - Klinicki odjel za vaskularnu kirurgiju, Split
  - University Hospital Dubrava, Zagreb
  - Zavod za vaskularnu kirurgiju, Zagreb
- Czechia (3):
  - Salvatella s.r.o., Třinec, Dolni Lomna
  - CHIR-Chirurgické oddeleni, Jihlava
  - U Nemocnice v Praze, Prague
- France (3):
  - Hopital Michallon, Grenoble, La Tronche
  - Hopital Nord Franche-Comte, Belfort, Trevenans
  - Hopital Rothschild - AP-HP, Paris, Île-de-France Region
- Germany (5):
  - Department od Dermatology, Venerology and Allergology, University of Essen, Essen, North Rhine-Westphalia
  - Gemeinschaftspraxis Drees.K.CH.Busch/v.d.Ecken, Dortmund
  - Technische Universitaet Dresden - Universitaetsklinikum Carl Gustav Carus - Klinik fuer Dermatologie, Dresden
  - University Hospital Erlangen, Erlangen
  - Oberhausen Sterkrade (Zweigpraxis), Oberhausen
- Hungary (6):
  - Bugat Pal Korhaz, Gyöngyös, Heves County
  - DermaMed Research Kft, Orosháza, Oroshaza
  - Clinexpert Kft, Budapest
  - Debreceni Egyetem, Klinikai Kozpont, Borgyogyaszati Klinika, Debrecen
  - Markhot Ferenc oktatókórház és rendelöintézet, Eger
  - BKS Research Kft, Hatvan
- Poland (5):
  - Uslugi Medyczne PRO-MED Sp. z.o.o, Gliwice, Gliwicie
  - Szpital Uniwersytecki nr 1 im. dr. A. Jurasza w Bydgoszczy Poradnia Leczenia Ran Przewleklych, Bydgoszcz
  - Nzoz Gam-Med, Kielce
  - MIKOMED Sp. Z.o.o., Lodz
  - Braci Wieniawskick 12B, Lublin
- United Kingdom (2):
  - Hull University Teaching Hospitals NHS Trust, Hull
  - Accelerate CIC, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Venous Leg Ulcer Standard of Care With Granulox: Subjects will receieve standard of care treatment with Granulox added as an adjunct therapy.
  Venous Leg Ulcer Standard of Care with Granulox: Granulox will be added as an adjunct therapy to defined standard of care in subjects with predominantly venous leg ulcers.
Period: Overall Study
Arm/Group | Venous Leg Ulcer Standard of Care | Venous Leg Ulcer Standard of Care With Granulox
Started | 66 | 62
Completed | 57 | 57
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Venous Leg Ulcer Standard of Care | Venous Leg Ulcer Standard of Care With Granulox | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (13) | 69.7 (10.4) | 70.25 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 33 | 68
  Male | 22 | 24 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 54 | 53 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  Hungary | 10 | 12 | 22
  Czechia | 2 | 3 | 5
  Poland | 36 | 37 | 73
  United Kingdom | 1 | 0 | 1
  France | 3 | 3 | 6
  Germany | 1 | 0 | 1
  Croatia | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Complete Wound Closure
Description: Confirmed Complete wound Closure is defined as an blinded assessment and observation of 100% re-epithelialization, confirmed by a second visit 15 days later (+/- 3 days).
Time Frame: Up to 20 weeks post therapy initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Leg Ulcer Standard of Care | Venous Leg Ulcer Standard of Care With Granulox
Number analyzed (Participants) | 57 | 57
Participants
  Yes | 11 | 9
  No | 46 | 48

ADVERSE EVENTS:
Time Frame: Up to 20 weeks post baseline
Description: Number of patients in Patient flow is calculated from FAS which had 114 patients. Participants at risk are taken from the safety population which is greater at 128 patients.
Arm/Group | Venous Leg Ulcer Standard of Care | Venous Leg Ulcer Standard of Care With Granulox
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/62
Serious Adverse Events (participants affected / at risk) | 3/66 | 2/62
Other Adverse Events (participants affected / at risk) | 6/66 | 7/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venous Leg Ulcer Standard of Care (N=66) | Venous Leg Ulcer Standard of Care With Granulox (N=62)
Inflammation of left leg (General disorders) | 0 (0) | 1 (1)
Stroke (thrombotic) (Vascular disorders) | 0 (0) | 1 (1)
Motor deficit of the lower limbs and mechanical fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shortness of breath (General disorders) | 1 (1) | 0 (0)
Worsening of coronary artery disease (acute myocardial infarction) (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venous Leg Ulcer Standard of Care (N=66) | Venous Leg Ulcer Standard of Care With Granulox (N=62)
Deterioration of basalioma on the face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Heart arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Inflammation of left leg (General disorders) | 0 (0) | 1 (1)
Flu syndrome (Infections and infestations) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Covid-19 infection (Infections and infestations) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Itching of the body (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT04181320/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT04181320/SAP_001.pdf